CLINICAL TRIAL: NCT02689947
Title: Evaluation of the Efficacy of Restylane Silk in the Correction of Tear Trough Deformity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nashville Centre for Laser and Facial Surgery (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Restylane Silk for Tear Trough
Record Dates: First submitted 2016-02-04; First posted 2016-02-24 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Tear Trough Deformity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restylane Silk (Experimental): open label no placebo control
  Interventions: Device: Restylane Silk

INTERVENTIONS:
Device: Restylane Silk

SUMMARY:
Prospective single center study to evaluate the safety and effectiveness of Restylane Silk for treatment of tear trough correction.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 21 and 65 years old
2. Tear trough deformity, Hirmand Type-1 and Type-2
3. Is voluntarily willing to consent to participate in the study
4. Is willing to comply with all requirements of the study including being photographed, follow post treatment care instructions, to attend all treatment, and follow up visits
5. Willingness to waive rights to use of still photos of themselves for research, marketing, or promotional reasons, including on the internet and on social media outlets.
6. Willingness to refrain from other surgical, laser, or injectable treatments in the periorbital region during the entire duration of the study.
7. Ability to provide informed consent.

Exclusion Criteria:

1. Marked delineation of the inferior orbital rim in the lateral aspect of the eyelid/orbit
2. Use of botulinum toxin in the periorbital region within the past 6 months.
3. Treatment with injectable fillers in the midface or periorbital region within the past 2 years or treatment at any time in the past with a permanent filler in the midface or periorbital region such as silicone, or PMMA (Artefill)
4. Laser skin resurfacing of the periorbital region within the past one year.
5. History of lower eyelid blepharoplasty or periorbital surgery in tear trough region.
6. The subject has a coagulation disorder or is currently using anti-coagulation medication
7. History of facial nerve palsy.
8. Inability to discontinue the use of nonsteroidal anti-inflammatory drugs or anticoagulants prior to treatment.
9. Current participation in another active clinical trial protocol
10. Presence of malar festoons
11. Active cutaneous infections
12. Allergy or sensitivity to benzocaine, lidocaine, prilocaine, or tetracaine.
13. Pregnant or nursing females
14. Other factors as deemed by the Principal Investigator that would make a subject unqualified for participation.
15. The subject has a history of keloids or compromised wound healing
16. The subject has a known adverse reaction to previous injection with hyaluronic acid or other subcutaneously injected device

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Primary outcome effectiveness analysis will test for the mean difference and overall improvement of radial smile lines based on baseline assessment and changes to the 6 month visit | baseline to month 6
  Primary outcome effectiveness analysis will test for the mean difference in improvement in terms of baseline to Month 6